CLINICAL TRIAL: NCT03604510
Title: Role of Frontal Cortex in the Pathophysiology of Gilles de la Tourette Syndrome (GTS)
Acronym: TIC-EEG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: CHUBX2016/41
Record Dates: First submitted 2018-04-05; First posted 2018-07-27 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Tourette Syndrome
MeSH Terms: conditions — Tourette Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Electroencephalographic recordings (Experimental): Electroencephalographic recordings
  Interventions: Procedure: Electroencephalographic recordings

INTERVENTIONS:
Procedure: Electroencephalographic recordings — 24 hours of electroencephalographic recordings (EEG-Holter) of prefrontal activity of Tourette's syndrome (TS) patients in ecological conditions.

SUMMARY:
Tourette's syndrome (TS) is a debilitating and severe syndrome whose pathophysiology remains unclear.

In order to precise the cortical regions involved in the generation of tics, investigators will realize an electroencephalogram (EEG) recording in the frontal cortex of TS patients in ecological conditions (EEG-holter). Activity changes will be correlated with event markers of tics and neurovegetative parameters. Statistical analyses will be compared between epochs of EEG recording with tics and without tics. The aim is to define the cortical regions involved in the genesis of tics in order to consider new targets for cortical stimulation.

DETAILED DESCRIPTION:
Gilles de la Tourette syndrome (GTS) is a childhood-onset disorder characterized by the presence of multiple motor tics and at least one vocal tic often associated with psychiatric co-morbidity. The expression of tics range from brief, recurrent and non-rhythmic motor or vocal actions (simple tics) to complex motor or vocal sequences (complex tics). The pathophysiology of tics is not yet fully understood. Recent imaging data suggest that the pattern of functional connectivity in cortico-basal ganglia networks is disrupted in GTS patients and could reflect a defect in brain maturation. However, regions involved in the immediate genesis of tics remains unknown since it is difficult to capture on line the cortical changes associated with tic generation using imaging techniques due to moving artefacts. Moreover, tics are much more frequent in everyday life conditions than in the artificial conditions of a laboratory. The aim is to study cortical activity changes occurring before tic occurrence by using long duration recording of encephalographic activity (EEG) in ecological conditions through Holter EEG techniques (24h recordings). Recordings will be performed in 15 patients with a severe form of Tourette's syndromes. EEG changes will be correlated to event markers, voluntary monitored by patients or automatically recorded (accelerometers for motor tics). EEG epoch centered on tics will be compared to similar epochs without tics. The occurrence of tics will also be correlated with neurovegetative markers of emotions such as RR interval ECG variability and skin resistivity changes. The ultimate goal of this project is to define a potential therapeutic target of tics for chronic cortical stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Tourette's syndrome since at least 2 years
* Lack of psychiatric comorbidity of axis 1 (depression)
* Y-YSGT score > 20
* Social insurance in accordance with the french law

Exclusion Criteria:

* Epilepsia
* Patient with an implanted medical device
* Severe mental or somatic disease
* Risk of suicide,
* Pregnant or breast feeding women
* Patient under "curatelle" or "tutelle"
* Patient hospitalized

no social insurance

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2018-02-02 (Actual); Primary Completion 2020-03-03 (Actual); Study Completion 2020-03-03 (Actual)

PRIMARY OUTCOMES:
Electroencephalogram (EEG) signal | During 24 hours
  24 hours recording of encephalographic activity (EEG) in ecological conditions through Holter EEG.

SECONDARY OUTCOMES:
Tic occurence | During 24 hours
  Occurence of tic recorded by the patient with a button press connected with a case and automatically recorded with an accelerometers for motor tics.
Age | Day 0
Gender | Day 0
Disease duration | Day 0
Neurovegetative marker of emotions : RR Interval | During 24 hours
  Intervals between R waves (RR interval) from the electrocardiogram
Neurovegetative marker of emotions : skin conductance | During 24 hours
  Skin conductance registered with a Bracelet sensor
MINI (Mini International Neuropsychiatric Interview) | Day 0
Montgomery and Asberg Depression Rating Sacle (MADRS) Score | Day 0
State Trait Anxiety Inventory (STAI A and B) | Day 0
Global Assessment of Functioning Score (Global Assessment of Functioning Scale) | Day 0
Yale Global Tic severity score (YGTS) | Day 0
ADHD RS rating score (ADHD RS rating Scale) | Day 0
Yale Brown Obsessive Compulsive Score (Y-BOCS Scale) | Day 0
Obsessive-Compulsive Inventory-Revised Score (OCI-R) | Day 0

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No